CLINICAL TRIAL: NCT01889303
Title: Phase II Clinical Trial of Docetaxel Plus Cisplatin as Adjuvant Chemotherapy and Concurrent Chemoradiotherapy Versus FOLFOX6 as Adjuvant and 5-FU/CF as Chemoradiotherapy in Patients of Locally Advanced Gastric Cancer After Radical Surgery
Brief Title: Phase II Study of DC Versus 5-FU/CF as Chemotherapy and Concurrent Chemoradiotherapy for Locally Advanced Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wuhan University (Other)
Responsible Party: Principal Investigator, Zhou Fuxiang, Deputy director of the department of Radiation and medical oncology, Wuhan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCCSC G-02
Record Dates: First submitted 2013-06-02; First posted 2013-06-28 (Estimated); Last update posted 2022-02-14 (Actual); Status verified 2022-01

CONDITIONS: Gastric Cancer
Keywords: concurrent chemoradiotherapy; FOLFOX6; chemotherapy; docetaxel; cisplatin; gastric cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Chemoradiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Active Comparator): chemotherapy regimen:Oxaliplatin 85mg/m2 IV d1,Leucovorin 400mg/m2 IV d1,5-FU 400mg/m2 IV bolus d1 ,then 2400mg/m2 over 46h continuous infusion Q2W for 3 cycles → 5-FU 400 mg/m2 IV and Leucovorin 20 mg/m2 IV on the first four and the last three days of radiotherapy + RT 45Gy (5weeks)→ Rest for 4 weeks →Oxaliplatin 85mg/m2 IV d1,Leucovorin 400mg/m2 IV d1,5-FU 400mg/m2 IV bolus d1 ,then 2400mg/m2 over 46h continuous infusion Q2W for 3 cycles.
  Radiation: concurrent chemoradiotherapy with 5-FU/CF.Radiotherapy consisted of 45Gy of radiation at 1.8Gy per day, five days per week for five weeks.
  Interventions: Drug: concurrent chemoradiotherapy with 5-FU/CF; Radiation: radiation
- Arm B (Experimental): chemotherapy regimen:Docetaxel 75mg iv D1,Cisplatin 75mg iv D1 ,Q3W x 2 cycles → Docetaxel 35mg iv D1,Cisplatin 25mg iv D1,QWx4 cycles(but rest in the 4th week during RT) + RT 45Gy (5weeks) for concurrent chemoradiotherapy→ Rest for 4 weeks → Docetaxel 75mg iv D1,Cisplatin 75mg iv D1 ,Q3W x 2 cycles
  Radiation: concurrent chemoradiotherapy with DC.Radiotherapy consisted of 45Gy of radiation at 1.8Gy per day, five days per week for five weeks.
  Interventions: Drug: DC; Radiation: radiation

INTERVENTIONS:
Drug: DC — Docetaxel plus cisplatin chemotherapy regimen was delivered as chemotherapy and concurrent chemoradiotherapy.
  chemotherapy regimen: Docetaxel（Qilu Pharma. China） 75mg iv D1, Cisplatin（Qilu Pharma. China） 75mg iv D1 ,Q3W for 2 cycles, then Docetaxel 35mg iv D1, Cisplatin 25mg iv D1,QWx4 cycles(but rest in the 4th week during RT) + RT 45Gy( 5weeks) for concurrent chemoradiotherapy→ Rest for 4 weeks → Docetaxel 75mg iv D1,Cisplatin 75mg iv D1 ,Q3W for 2 cycles.
  Other Names: Docetaxel Injection， Hengrui Medicine
  Arms: Arm B
Drug: concurrent chemoradiotherapy with 5-FU/CF — FOLFOX6 regiment was delivered as adjuvant chemotherapy and 5-FU/CF as concurrent chemotherapy treatment.
  Adjuvant chemotherapy: FOLFOX6 regiment : Oxaliplatin（Hengrui Medicine Co., Ltd，China） 85mg/m2 IV d1, Leucovorin （Hengrui Medicine Co., Ltd，China）400mg/m2 IV d1, 5-FU（Hengrui Medicine Co., Ltd，China） 400mg/m2 IV bolus d1, followed with 2400mg/m2 over 46h continuous infusion Q2Wx3 cycles of chemotherapy Concurrent chemotherapy : 5-FU 400mg/m2 IV and Leucovorin 20mg/m2 IV were given on the first four and the last three days in the period of radiotherapy. After radiation, patients will have a rest lasting for 4 weeks and then given Folxof6 regiment chemotherapy for 3 cycles.
  Other Names: Hengrui Medicine
  Arms: Arm A
Radiation: radiation — Therapy plan system was formulated by CT simulation. Radiation was delivered with 15MV photons in both Arm A and Arm B. Radiotherapy consisted of 45Gy of radiation at 1.8Gy/day, five days per week for 5 weeks, to the tumor bed, to the margins of resection, to the regional nodes. Protection of spinal cord, heart, liver and kidney should be considered.

SUMMARY:
Concurrent chemoradiotherapy has been demonstrated a significant improvement in overall survival and disease-free survival according to Intergroup Trial 0116 in patients with gastric cancer after surgical resection. However,there are still many patients experiencing local recurrence or distant metastasis after adjuvant chemotherapy and concurrent chemoradiotherapy for locally advanced gastric cancer after resection. The optimal and standard regimen for adjuvant treatment has not been established in locally advanced gastric cancer yet.The investigators designed the trial to investigate the efficacy and safety of docetaxel plus cisplatin regimen as adjuvant chemotherapy and concurrent chemoradiotherapy regimen compared with classical FOLFOX6 regimen as adjuvant chemotherapy and 5-FU/CF as chemoradiotherapy in patients of locally advanced gastric cancer after D2 radical resection.

DETAILED DESCRIPTION:
In Intergroup 0116 trial, 5-FU plus CF regimen was used as adjuvant chemotherapy and concurrent chemoradiotherapy in patients with resected gastric cancer.But 33 percent of those in the chemoradiotherapy group had distant relapses. Docetaxel plus cisplatin regimen as adjuvant chemotherapy for gastric cancer has been proofed Safe and Effective in many clinical trials about gastric cancer. The purpose of this study is to evaluate efficacy and safety of docetaxel plus cisplatin regimen as adjuvant chemotherapy and concurrent chemoradiotherapy regimen compared with classical FOLFOX6 regimen as adjuvant chemotherapy and 5-FU/CF as chemoradiotherapy in patients of locally advanced gastric cancer after D2 radical surgery. The investigators hope the new interventions can reduce the rate of distant metastasis and have more clinical benefit.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Age > 19
3. Histologically proven gastric or gastroesophageal adenocarcinoma
4. ≥ D2 lymph node dissection, curative gastrectomy,
5. Stage T4 with or without any positive LN (AJCC 2010) ，No distant metastasis(M0) and after D2 radical gastrectomy
6. KPS≥70 or ECOG 0-2
7. R0 resection,
8. Adequate bone marrow functions (WBC≥4.0×109/L，GRAN≥2.0×109/L，Hb≥90g/L, transfusion allowed, PLT≥100×109/L )
9. No severe functional damage of major organ,and no uncontrolled or severe cardiopulmonary concurrent system disease
10. Adequate renal functions(serum creatinine ≤ 1.5×ULN ) ;liver functions (serum bilirubin ≤ 1.5×ULN, AST/ALT ≤ 2.5 times(normal value) ,serum AKP≤2.5×ULN
11. Predictive survival time longer than 6 months.

Exclusion Criteria:

1. pregnant or breast-feeding women;
2. Have received preoperative neoadjuvant therapy of gastric cancer
3. Before or at the same time with other malignant tumor, and underwent chemotherapy, immune, and biological treatment and radiation therapy;with the exception of adequately treated cervical carcinoma in situ or localized non-melanoma skin cancer
4. uncontrolled mental disease
5. Severe or uncontrolled cardiovascular disease (congestive heart failure NYHA III or IV, no myocardial infarction within the last 12 months, unstable angina pectoris, or significant arrhythmia)
6. Active infection requiring antibiotics
7. Resection margin (+) at permanent pathology
8. Peripheral neuropathy symptoms, NCI class > 1
9. severe malnutrition or severe anemia
10. uncontrolled Primary brain tumors or the central nervous system disease
11. Known hypersensitivity against any of the study drugs
12. Pathologic stage I-IIa or IV (according to AJCC 2010)
13. Inadequate surgery including D0, D1 resection, dissected LNs less than 12
14. Concurrent treatment with other experimental drugs or other anti-cancer therapy, or treatment within a clinical trial within 30 days prior to trial entry

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-05; Primary Completion 2023-06-01 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | 2,3 year
  efficacy of docetaxel plus cisplatin regimen as adjuvant chemotherapy and concurrent chemoradiotherapy for locally advanced gastric cancer patients in this trial is defined as 2 or 3 year disease free survival

SECONDARY OUTCOMES:
Overall survival(OS) | 3 year
  efficacy of docetaxel plus cisplatin regimen as adjuvant chemotherapy and concurrent chemoradiotherapy for locally advanced gastric cancer patients in this trial is defined as 3-year overall survival
Local and regional control rate | 2,3 year
  efficacy of docetaxel plus cisplatin regimen as adjuvant chemotherapy and concurrent chemoradiotherapy for locally advanced gastric cancer patients in this trial is defined as local and regional control rate
feasibility (including adverse events ) | 3year
  feasibility of docetaxel plus cisplatin regimen as adjuvant chemotherapy and concurrent chemoradiotherapy for locally advanced gastric cancer patients in this trial is defined as toxicities and rate of patients complete concurrent chemoradiation according to protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Y F Zhou, PHD, Principal Investigator — President of Zhongnan Hospital of Wuhan University
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided